CLINICAL TRIAL: NCT07266870
Title: The Effect of CORE on Nursing Students' Knowledge and Attitude Levels Regarding Pain Assessment: Randomized Controlled Trial
Brief Title: Effect of CORE on Knowledge and Attitude Levels Regarding Pain Assessment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Müjgan ONARICI, Asst. Prof., Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CAKÜ
Record Dates: First submitted 2025-11-17; First posted 2025-12-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Nursing Education
Keywords: CORE; Pain assessment; Nursing education; Attitude; Knowledge
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: The study will be conducted using a randomised controlled experimental design.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CORE application (Experimental): During the study implementation process, a knowledge test and attitude scale will be administered as a pretest, posttest, and retention test. Case scenarios prepared for pain assessment will be applied to the intervention group students as CORE application.
  Interventions: Behavioral: CORE application
- Control (No Intervention): During the study implementation process, a knowledge test and attitude scale will be administered as a pretest, posttest, and retention test.

INTERVENTIONS:
Behavioral: CORE application — Case scenarios prepared for pain assessment will be applied to the intervention group students as CORE application.
  Arms: CORE application

SUMMARY:
CORE is an assessment tool that uses written scenarios designed to address problems that students may encounter in real clinical settings. These scenarios are presented at different stations. It enables educators to conduct more objective evaluations during the learning process, contributing to effective learning by providing students with immediate feedback. This research will examine the effect of CORE on nursing students' knowledge and attitudes regarding pain assessment. The study will be conducted using a randomised controlled experimental design. The study population will consist of senior nursing students taking the Nursing Professional Practice II course in the spring semester of the 2025/26 academic year at a nursing department in the Central Anatolia region of Turkey (n = 100). The sample for the study will consist of students who agree to participate in the research. Students will be randomized into intervention and control groups based on their pre-test knowledge scores. Research data will be collected using the "Personal Information Form" "Pain Knowledge Test", "Nursing Students' Attitudes Scale Toward Pain Assessment" and "CORE Satisfaction Form". Approval from the ethical committee has been obtained for the research to be conducted, and written permission has been requested from the institution in which the research will take place. Before starting the research, students will be informed about it and asked to provide written informed consent. Students in the intervention group will perform the CORE application on tablets using case scenarios prepared for pain assessment in the Nursing Skills Laboratory. Data collection tools will be administered three times: pre-test, post-test, and retention test. Only the "CORE Satisfaction Form" will be administered to students in the intervention group to assess their satisfaction after the CORE application. Descriptive statistics and the Student's t-test, Mann-Whitney U-test, t-test and Wilcoxon signed-rank test for dependent groups will be used in the analysis of the data.

DETAILED DESCRIPTION:
Study procedure:

* Research data will be collected from students enrolled on the Practice II course of the Nursing Profession programme during the spring semester of the 2025/26 academic year. The following tests and questionnaires will be administered as pre-tests before the topic is explained during the first week of the semester's face-to-face theoretical training:

  * A "Personal Information Form"
  * A "Pain Knowledge Test"
  * The "Nursing Students' Attitudes Toward Pain Assessment Scale" Pain and CORE training will then be provided.
* Before the study begins, students will be informed about it and their written informed consent will be obtained.
* The intervention and control groups will be randomised based on their pre-test knowledge scores using www.randomizer.org.

Following randomisation, intervention group students will use the CORE application on a tablet with case scenarios prepared for pain assessment in the Nursing Skills Laboratory on the fifth day after theoretical training.

One day after implementation, both groups will take the 'Pain Knowledge Test' and the 'Nursing Students' Attitudes Towards Pain Assessment Scale' again, this time as a post-test. The 'CORE Satisfaction Form' will be given to the intervention group to measure their satisfaction with the CORE experience.

• Two weeks after the CORE implementation, both groups will take the 'Pain Knowledge Test' and the 'Nursing Students' Attitudes Towards Pain Assessment Scale' again, this time as a retention test to assess knowledge retention and attitude levels.

After the data collection phase of the study is complete, CORE will also be administered to the control group.

• Before implementation, a pilot study will be conducted with five students from outside the target group to assess the clarity of the data collection forms and the length of the CORE scenarios.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in research
* Taking the Nursing Professional Courses Practicum II course
* Participating in pain education
* Participating in CORE training

Exclusion Criteria:

* Not attending training
* Not completing data collection tools

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — All
Enrollment: 100 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2026-02-18 (Estimated); Study Completion 2026-03-09 (Estimated)

PRIMARY OUTCOMES:
1. Differences of knowledge scores between groups | To assess their knowledge levels, the pretest was administered in the first week, the posttest in the second week (1 day after the CORE application), and the retention test in the fourth week. Total duration: 4 weeks.
  Pre-test, post-test and retention tests were applied to measure the level of knowledge. The 'Pain Knowledge Test', which was prepared by the researchers, will be used to assess knowledge levels. The test consists of ten questions. It will be marked out of 100. Test scores obtained at three different times will be compared. Higher post-test and retention test scores than pre-test scores suggest an increase in knowledge.

SECONDARY OUTCOMES:
Differences in Attitude Scores Towards Pain Assessment Between Groups | To assess attitudes, a pre-test was administered in the first week, a post-test in the second week (1 day after the CORE application), and a retention test in the fourth week. Total duration: 4 weeks.
  Pre-test, post-test and retention tests were applied to measure attitudes. The "Nursing Students' Attitudes Scale Toward Pain Assessment" scale will be used to evaluate students' attitudes towards pain assessment. The scale consists of 15 items and two subfactors. Factor 1 represents the importance of pain assessment, while Factor 2 represents the interest subscale. The minimum possible score is 15, and the maximum possible score is 75. As the scale score increases, so do nursing students' positive attitudes towards pain assessment.

CONTACTS AND LOCATIONS:
Overall Officials: MÜJGAN ONARICI, PhD, Principal Investigator — Çankırı Karatekin University

IPD SHARING:
Plan to Share IPD: No
in progress

REFERENCES:
- [Background] Madenoğlu Kıvanç, M., Türen, S., Gül, A., Turan Miral, M., Atakoğlu Yılmaz, R., & Kara Özçalık, C. (2023). Hemşirelik eğitiminde öğrenci değerlendirme stratejisi: Objektif yapılandırılmış klinik sınavı. Sağlık ve Yaşam Bilimleri Dergisi, 5(2), 80-86. DOI: 10.33308/2687248X.202352301.
- [Background] Hakbilen HG, Ince S. Effect of Kegel Exercise-Focused Intervention on Urinary Incontinence in Elderly Women. J Wound Ostomy Continence Nurs. 2025 Mar-Apr 01;52(2):137-146. doi: 10.1097/WON.0000000000001162. Epub 2025 Mar 20. PMID 40136104
- [Background] Turhan, K., Unsal, S., Kalaycı, N., Kayıkçı, V., & Uzun, E. (2006). Computer supported clinically oriented reasoning exam management system with client/server architecture: CORE-Builder. Current Developments in Technology-Assisted Education, 1203-1207.